CLINICAL TRIAL: NCT01245621
Title: Early vs. Later Palliative Cancer Care: Clinical and Biobehavioral Outcomes
Brief Title: Study of Palliative Care Intervention for Advanced Cancer Patients and Their Caregivers -Educate Nurture Advise Before Life Ends (ENABLE III)
Acronym: ENABLE III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NCCC-BAKI: D0946; R01NR011871-01 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-22 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Cancer
Keywords: palliative care; end of life care; quality of life; caregivers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early entry group (Active Comparator): Early entry group will begin the intervention at time of diagnosis of advanced cancer
  Interventions: Behavioral: Early palliative care intervention
- Later entry group (Active Comparator): Later entry group will begin the intervention 12 weeks after enrollment in the study.
  Interventions: Behavioral: Later entry group

INTERVENTIONS:
Behavioral: Later entry group — 1. Advanced Practice Palliative Care Nurse Interventionist instituting a phone-based: a) Charting Your Course (CYC)-Patient Curriculum (6-session manualized); b) Creativity Optimism Planning Expert Information (COPE) Caregiver Curriculum (3 session manualized) and c) ongoing contact as determined by the Palliative Care Team assessment/plan; and
  2. Comprehensive Palliative Care Team Assessment & Management Plan.
  Arms: Later entry group
Behavioral: Early palliative care intervention — 1. Advanced Practice Palliative Care Nurse Interventionist instituting a phone-based: a) Charting Your Course (CYC)-Patient Curriculum (6-session manualized); b) Creativity Optimism Planning Expert information(COPE) Caregiver Curriculum (3 session manualized) and c) ongoing contact as determined by the Palliative Care Team assessment/plan; and
  2. Comprehensive Palliative Care Team Assessment & Management Plan.
  Arms: Early entry group

SUMMARY:
ENABLE III is a randomized clinical trial that evaluates a phone-based palliative care intervention designed to improve quality of life, mood, and symptom management for patients with an advanced stage cancer and their caregivers.

The primary aims of this clinical trial are to determine whether a palliative care intervention (introduced immediately or 12 weeks after diagnosis) can improve survival, quality of life, mood, symptom intensity and end-of-life care.

DETAILED DESCRIPTION:
In 2008, cancer claimed more than 565,000 American lives -1,500 people a day. Palliative care strives to improve quality of life (QOL) and to prevent "bad deaths" by providing expert, interdisciplinary care to manage the effects of disease and treatment. Effective end-of-life (EOL) care depends upon proactive, patient-centered interventions to prepare patients and families for the challenges of terminal illness. We were able to demonstrate the feasibility and efficacy of a concurrent oncology palliative care (COPC) intervention in improving quality of life and mood in our previous studies ENABLE I and ENABLE II; however, a number of gaps in our knowledge remain.

Patients will be randomized to begin the intervention either immediately or 12 weeks after a new diagnosis of advanced or recurrent cancer. This phone-based intervention consists of: 1) an Advanced Practice Palliative Care Nurse Interventionist instituting 1a) a 6-session manualized patient curriculum- Charting Your Course (CYC), 1b) a 3-session manualized, caregiver curriculum- the Creativity Optimism Planning Expert information (COPE) program, and 1c) on-going patient and caregiver follow up; and 2) Palliative Care Team Comprehensive Assessment & Management.

ELIGIBILITY:
INCLUSION CRITERIA FOR PATIENTS:

1. Able to speak and understand English
2. Over age 18
3. NEW diagnosis, recurrence, or progression of an advanced stage cancer within THIRTY days of the date the patient was informed of the diagnosis by his/her oncology clinician.
4. Estimated survival of 2 years or less
5. Diagnosed with an advanced stage cancer such as one of the following:

   * Lung Cancer: Stage IIIB or IV non-small cell, or extensive stage small cell
   * Breast Cancer: Stage IV with poor prognostic indicators including but not limited to: a) >2 cytotoxic regimens for MBC; b) diagnosis of MBC less then or equal to 12 months since completion of adjuvant or neoadjuvant treatment; c) triple negative disease (ER/PR - and Her 2-);d) parenchymal brain mets and/or carcinomatous meningitis
   * Gastrointestinal (GI) Cancers: Unresectable stage III or IV
   * Genitourinary (GU) Cancers: Stage IV (for prostate cancer inclusion is limited to persons with hormone refractory prostate cancer)
   * Brain Cancer: Unresectable, Grade IV
   * Melanoma, Stage IV
   * Hematologic Malignancies -Leukemia (e.g. acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myeloid leukemia (CML), chronic lymphocytic leukemia (CLL) - advanced stage, treatment refractory, poor prognosis cell type or chromosomal abnormalities, "older age" -Lymphoma- Stage IV or treatment refractory Hodgkin's disease or non-Hodgkin's lymphoma -Multiple Myeloma - elevated β2-microglobulin, albumin <3.5, PCLI >1%, CRP >6µg/mL, elevated LDH, plasmablastic morphology, abnormal. chromosome 13.
6. Completion of baseline interview

INCLUSION CRITERIA FOR PATIENTS FOR BIOMARKER SUB-STUDY:

1. Only patients with lung, breast, GI, GU cancer are eligible

INCLUSION CRITERIA FOR CAREGIVERS:

1. Able to read and understand English
2. Anyone identified by the patient as "a person who knows you well & is involved in your medical care".

PATIENT EXCLUSION CRITERIA:

1. Dementia or significant confusion (Impaired cognitive status as indicated by a score of 3 or less on the Callahan six-item cognitive screening tool 18)
2. Axis I psychiatric diagnosis of severe mental illness (DSM-IV) (e.g. schizophrenia, bipolar disorder, or active substance use disorder)
3. Patients will not be excluded if they do not identify a caregiver
4. Prior involvement with palliative care service within the last year
5. Minimum predicted survival of less than 12 weeks (3 months)

PATIENT BIOMARKER SUBSTUDY EXCLUSION CRITERIA:

1. Receiving chronic steroid hormones or unable to schedule specimen collection distant from chemotherapy from steroid pre-medications
2. Unable to come to Norris Cotton Cancer Center (NCCC) for specimen collection times.

CAREGIVER EXCLUSION CRITERIA:

1. Unwilling to participate in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in patient's quality of living over time | baseline, 6,12,18,24,36 and every 12 weeks until death or end of study
  Quality of living assessments will include quality of life (QOL), mood, and symptom intensity measures using the following measures:
  * Functional Assessment of Chronic Illness Therapy-Palliative Care (FACIT-Pal):
  * Quality of Life at End of Life (QUAL-E).
  * Center for Epidemiological Study- Depression (CES-D).
Quality of end of life care | chart review at time of death and caregiver proxy interview 2-3 months after patient death
  End of life (EOL) Care Data Collection Form: This form is used to collect information about the quality of EOL care and circumstances surrounding the last 48 hours of life for patients who die in hospital, nursing home, or home.
  Quality of Dying and Death Measure (QODD). The QODD is a structured interview conducted with a caregiver to measure the quality of a patient's last week of life. The interview assesses the caregiver's perception of patient symptoms, preferences, and satisfaction with care.
Estimate and compare the hazard ratios and median survival before and after 1 year from enrollment | From enrollment until patient death or end of study
  We hypothesize that Early entry patients will have longer overall survival at one year compared with Later entry patients.
Change in caregiver quality of life, burden and grief over time | baseline, 6,12,18,24,36, and every 12 weeks until patient death or end of study
  Caregiver burden and QOL will be measured using:
  * Quality of Life- Cancer- a self-report measure of QOL for caregivers of patients with cancer.
  * Montgomery Borgatta Caregiver Burden Scale -a self-report measure of caregiver burden.
  * Center for Epidemiological Study- Depression CESD is a measure of depressive symptoms.
  * Functional Assessment of Chronic Illness Therapy - Spiritual Module (FACIT-Sp) - a measure of spiritual well-being developed for persons with chronic illness.
  * Prigerson Inventory of Complicated Grief-Short form (ICG-SF) embedded in the Quality of Death and Dying (QODD).

SECONDARY OUTCOMES:
Mediating mechanisms and moderators of the concurrent palliative care intervention. | baseline, 6,12,18,24,36 weeks and every 12 weeks until death or end of study
  Mediating mechanisms measured will include patient activation, decision support, goal setting, problem solving, care coordination.
  Moderators measures will include: decision control and treatment goals, self-efficacy, optimism, coping style, social support.
Determine feasibility of enrolling less common solid tumors and hematologic malignancies. | Estimated recruitment period of 2 years
  ENABLE II recruited patients only with lung, breast, GI, and GU tumors. We will attempt to also recruit patients with less common "poor prognosis" solid tumors (e.g. brain) and hematologic malignancies and their caregivers for this concurrent oncology palliative care intervention.
Explore patterns of stress (diurnal salivary and plasma cortisol) and immune biomarkers (lymphocyte subsets and cytokines) | Baseline, 12, and 24 weeks
  We will explore patterns of stress (diurnal salivary and plasma cortisol) and immune biomarkers (lymphocyte subsets and cytokines)at baseline, 12, and 24 weeks after intervention in a subset of 50 patients with breast, lung, GI, and GU cancer.
  We hypothesize that stabilized or improved biomarkers of stress and immune function will be evident after Early and Later entry intervention participation.
Examine the relations among quality of life, mood, symptoms, survival, stress and immune biomarkers. | Baseline, 12, and 24 weeks
  We hypothesize that higher quality of life,mood, lower symptom intensity, and longer survival will be associated with stable or improved stress and immune biomarkers (e.g. normal plasma cortisol and diurnal salivary cortisol variability, lymphocyte subsets and cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Bakitas, DNSc, APRN, Principal Investigator — Dartmouth-Hitchcock Medical Center; Jennifer P. Frost, RN, MS, Study Director — Dartmouth-Hitchcock Medical Center
Locations (7):
- United States (7):
  - Dartmouth-Hitchcock Medical Center - Lebanon, Lebanon, New Hampshire
  - Dartmouth-Hitchcock Clinic - Manchester, Manchester, New Hampshire
  - St. Joseph Hospital, Nashua, New Hampshire
  - Dartmouth-Hitchcock NCCC Nashua, Nashua, New Hampshire
  - Providence VA Medical Center, Providence, Rhode Island
  - Mountainview Medical, Berlin Corners, Vermont
  - Veteran's Administration Hospital, White River Junction, Vermont

REFERENCES:
- [Background] O'Hara RE, Hull JG, Lyons KD, Bakitas M, Hegel MT, Li Z, Ahles TA. Impact on caregiver burden of a patient-focused palliative care intervention for patients with advanced cancer. Palliat Support Care. 2010 Dec;8(4):395-404. doi: 10.1017/S1478951510000258. Epub 2010 Sep 28. PMID 20875202
- [Background] Bakitas M, Stevens M, Ahles T, Kirn M, Skalla K, Kane N, Greenberg ER; Project Enable Co-Investigators. Project ENABLE: a palliative care demonstration project for advanced cancer patients in three settings. J Palliat Med. 2004 Apr;7(2):363-72. doi: 10.1089/109662104773709530. PMID 15130218
- [Background] Bakitas M, Ahles TA, Skalla K, Brokaw FC, Byock I, Hanscom B, Lyons KD, Hegel MT; ENABLE project team. Proxy perspectives regarding end-of-life care for persons with cancer. Cancer. 2008 Apr 15;112(8):1854-61. doi: 10.1002/cncr.23381. PMID 18306393
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Barnett KN, Brokaw FC, Byock IR, Hull JG, Li Z, McKinstry E, Seville JL, Ahles TA. The project ENABLE II randomized controlled trial to improve palliative care for rural patients with advanced cancer: baseline findings, methodological challenges, and solutions. Palliat Support Care. 2009 Mar;7(1):75-86. doi: 10.1017/S1478951509000108. PMID 19619377
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Lyons KD, Bakitas M, Hegel MT, Hanscom B, Hull J, Ahles TA. Reliability and validity of the Functional Assessment of Chronic Illness Therapy-Palliative care (FACIT-Pal) scale. J Pain Symptom Manage. 2009 Jan;37(1):23-32. doi: 10.1016/j.jpainsymman.2007.12.015. Epub 2008 May 27. PMID 18504093
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Corn BW, Feldman DB, Hull JG, O'Rourke MA, Bakitas MA. Dispositional hope as a potential outcome parameter among patients with advanced malignancy: An analysis of the ENABLE database. Cancer. 2022 Jan 15;128(2):401-409. doi: 10.1002/cncr.33907. Epub 2021 Oct 6. PMID 34613617
- [Derived] Prescott AT, Hull JG, Dionne-Odom JN, Tosteson TD, Lyons KD, Li Z, Li Z, Dragnev KH, Hegel MT, Steinhauser KE, Ahles TA, Bakitas MA. The role of a palliative care intervention in moderating the relationship between depression and survival among individuals with advanced cancer. Health Psychol. 2017 Dec;36(12):1140-1146. doi: 10.1037/hea0000544. Epub 2017 Oct 19. PMID 29048177
- [Derived] Bagcivan G, Dionne-Odom JN, Frost J, Plunkett M, Stephens LA, Bishop P, Taylor RA, Li Z, Tucker R, Bakitas M. What happens during early outpatient palliative care consultations for persons with newly diagnosed advanced cancer? A qualitative analysis of provider documentation. Palliat Med. 2018 Jan;32(1):59-68. doi: 10.1177/0269216317733381. Epub 2017 Sep 27. PMID 28952887
- [Derived] Bakitas MA, Tosteson TD, Li Z, Lyons KD, Hull JG, Li Z, Dionne-Odom JN, Frost J, Dragnev KH, Hegel MT, Azuero A, Ahles TA. Early Versus Delayed Initiation of Concurrent Palliative Oncology Care: Patient Outcomes in the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1438-45. doi: 10.1200/JCO.2014.58.6362. Epub 2015 Mar 23. PMID 25800768
- [Derived] Dionne-Odom JN, Azuero A, Lyons KD, Hull JG, Tosteson T, Li Z, Li Z, Frost J, Dragnev KH, Akyar I, Hegel MT, Bakitas MA. Benefits of Early Versus Delayed Palliative Care to Informal Family Caregivers of Patients With Advanced Cancer: Outcomes From the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1446-52. doi: 10.1200/JCO.2014.58.7824. Epub 2015 Mar 23. PMID 25800762
- See also: Dartmouth-Hitchcock Norris Cotton Cancer Center home page — http://cancer.dartmouth.edu/